CLINICAL TRIAL: NCT00647088
Title: Genetic of Aortic Valve Stenosis - Clinical and Therapeutic Implications
Acronym: GENERAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: P070141
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2016-02

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic Valve stenosis; Genetic; Mineralisation inhibitors
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples DNA Tissue valve
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- aortic stenosis: various age and disease severity
- Controls: Controls free of valvular disease

SUMMARY:
Pathophysiology of Aortic Valve Stenosis remains poorly known. The aim of the present study is to identify genetic factors involved in this disease using a case control trial design.

DETAILED DESCRIPTION:
Aortic valve stenosis (AS) is the most common valvular disease and the second most common indication for cardiac surgery in Western countries. AS has long been considered as a passive and degenerative process. Recent data challenged this concept, showing that AS is an active and highly regulated process with some similarities to atherosclerosis. However, pathophysiology of AS remains poorly understood and preliminary data suggest that genetic factors may be involved. The aim of the present study is to identify genetic factors involved in this disease using a case control trial design (1000 patients with AS and 1500 controls with no evidence of valve disease). For all patients and controls, blood samples including DNA and echocardiography will be performed.

ELIGIBILITY:
Patients:

Inclusion criteria :

* Age >=18 years
* Pure isolated degenerative aortic valve stenosis

Exclusion criteria :

* Rheumatic, congenital or post-radiation aortic stenosis
* Severe renal insufficiency (clearance < 30 ml/min)
* Aortic insufficiency > or = grade 2/4
* Other valve disease > or = grade 2/4

Controls

Inclusion criteria :

- Age >=18 years

Exclusion criteria :

* Known first degree relative with aortic valve stenosis
* Severe renal insufficiency (clearance < 30 ml/min)
* Any valve disease > or = grade 2/4

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: case control study Case = patients with aortic valve stenosis Controls = participants free of aortic valve stenosis
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Estimated)
Dates: Start 2008-03; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Identification of genetic polymorphisms of fetuin-A, matrix-GLA protein, vitamin D receptor | end of the study

SECONDARY OUTCOMES:
Identification of other genetic polymorphisms | End of the Study

CONTACTS AND LOCATIONS:
Overall Officials: David Messika-Zeitoun, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Assistance Publique - Hôpitaux de Paris, Bichat Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perrot N, Theriault S, Dina C, Chen HY, Boekholdt SM, Rigade S, Despres AA, Poulin A, Capoulade R, Le Tourneau T, Messika-Zeitoun D, Trottier M, Tessier M, Guimond J, Nadeau M, Engert JC, Khaw KT, Wareham NJ, Dweck MR, Mathieu P, Pibarot P, Schott JJ, Thanassoulis G, Clavel MA, Bosse Y, Arsenault BJ. Genetic Variation in LPA, Calcific Aortic Valve Stenosis in Patients Undergoing Cardiac Surgery, and Familial Risk of Aortic Valve Microcalcification. JAMA Cardiol. 2019 Jul 1;4(7):620-627. doi: 10.1001/jamacardio.2019.1581. PMID 31141105
- [Derived] Pawade T, Clavel MA, Tribouilloy C, Dreyfus J, Mathieu T, Tastet L, Renard C, Gun M, Jenkins WSA, Macron L, Sechrist JW, Lacomis JM, Nguyen V, Galian Gay L, Cuellar Calabria H, Ntalas I, Cartlidge TRG, Prendergast B, Rajani R, Evangelista A, Cavalcante JL, Newby DE, Pibarot P, Messika Zeitoun D, Dweck MR. Computed Tomography Aortic Valve Calcium Scoring in Patients With Aortic Stenosis. Circ Cardiovasc Imaging. 2018 Mar;11(3):e007146. doi: 10.1161/CIRCIMAGING.117.007146. PMID 29555836
- [Derived] Kubota N, David Messika-Zeitoun D. P650Influence of fetunin-a level on progression of calcific aortic valve stenosis The COFRASA - GENERAC Study. Eur Heart J Cardiovasc Imaging. 2016 Dec 1;17(suppl_2):ii130-ii136. doi: 10.1093/ehjci/jew250.001. PMID 28415102
- [Derived] Arangalage D, Nguyen V, Robert T, Melissopoulou M, Mathieu T, Estellat C, Codogno I, Huart V, Duval X, Cimadevilla C, Vahanian A, Dehoux M, Messika-Zeitoun D. Determinants and prognostic value of Galectin-3 in patients with aortic valve stenosis. Heart. 2016 Jun 1;102(11):862-8. doi: 10.1136/heartjnl-2015-308873. Epub 2016 Feb 19. PMID 26896466
- [Derived] Guauque-Olarte S, Messika-Zeitoun D, Droit A, Lamontagne M, Tremblay-Marchand J, Lavoie-Charland E, Gaudreault N, Arsenault BJ, Dube MP, Tardif JC, Body SC, Seidman JG, Boileau C, Mathieu P, Pibarot P, Bosse Y. Calcium Signaling Pathway Genes RUNX2 and CACNA1C Are Associated With Calcific Aortic Valve Disease. Circ Cardiovasc Genet. 2015 Dec;8(6):812-22. doi: 10.1161/CIRCGENETICS.115.001145. Epub 2015 Nov 9. PMID 26553695
- [Derived] Chin CW, Messika-Zeitoun D, Shah AS, Lefevre G, Bailleul S, Yeung EN, Koo M, Mirsadraee S, Mathieu T, Semple SI, Mills NL, Vahanian A, Newby DE, Dweck MR. A clinical risk score of myocardial fibrosis predicts adverse outcomes in aortic stenosis. Eur Heart J. 2016 Feb 21;37(8):713-23. doi: 10.1093/eurheartj/ehv525. Epub 2015 Oct 21. PMID 26491110
- [Derived] Dreyfus J, Durand-Viel G, Raffoul R, Alkhoder S, Hvass U, Radu C, Al-Attar N, Ghodbhane W, Attias D, Nataf P, Vahanian A, Messika-Zeitoun D. Comparison of 2-Dimensional, 3-Dimensional, and Surgical Measurements of the Tricuspid Annulus Size: Clinical Implications. Circ Cardiovasc Imaging. 2015 Jul;8(7):e003241. doi: 10.1161/CIRCIMAGING.114.003241. PMID 26156015
- [Derived] Nguyen V, Cimadevilla C, Estellat C, Codogno I, Huart V, Benessiano J, Duval X, Pibarot P, Clavel MA, Enriquez-Sarano M, Vahanian A, Messika-Zeitoun D. Haemodynamic and anatomic progression of aortic stenosis. Heart. 2015 Jun;101(12):943-7. doi: 10.1136/heartjnl-2014-307154. Epub 2015 Feb 5. PMID 25655063
- [Derived] Kochtebane N, Passefort S, Choqueux C, Ainoun F, Achour L, Michel JB, Back M, Jacob MP. Release of leukotriene B4, transforming growth factor-beta1 and microparticles in relation to aortic valve calcification. J Heart Valve Dis. 2013 Nov;22(6):782-8. PMID 24597398
- [Derived] Cimadevilla C, Cueff C, Hekimian G, Dehoux M, Lepage L, Iung B, Duval X, Huart V, Tubach F, Vahanian A, Messika-Zeitoun D. Prognostic value of B-type natriuretic peptide in elderly patients with aortic valve stenosis: the COFRASA-GENERAC study. Heart. 2013 Apr;99(7):461-7. doi: 10.1136/heartjnl-2012-303284. Epub 2013 Jan 24. PMID 23349346